CLINICAL TRIAL: NCT05906862
Title: First-in-Human, Phase 1 Study of AMT-253, in Patients With Advanced Solid Tumors
Brief Title: AMT-253 in Patients With Selected Advanced Solid Tumours
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Multitude Therapeutics (Australia) Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Multitude Therapeutics Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT-253-01
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AMT-253 Dose Escalation (Experimental)
  Interventions: Drug: AMT-253

INTERVENTIONS:
Drug: AMT-253 — Administered intravenously

SUMMARY:
This first-in-human study will evaluate the Maximum Tolerated Dose (MTD) / the Recommended Phase 2 Dose (RP2D), safety, tolerability, anti-tumor activity, pharmacokinetics, pharmacodynamics and immunogenicity of AMT-253, in Patients with Advanced Solid Tumors

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be willing and able to sign the ICF, and to adhere to the study visit schedule and other protocol requirements.
* Age ≥18 years (at the time consent is obtained).
* Patients who have undergone at least one systemic therapy and have radiologically or clinically determined progressive disease during or after most recent line of therapy, and for whom no further standard therapy is available, or who are intolerable to standard therapy.
* Patients must have at least one measurable lesion as per RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy ≥ 3 months.
* Patients must have adequate organ function.
* Women of child bearing potential (WCBP), defined as a sexually mature woman who has not undergone surgical sterilization or who has not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months) must agree to use two effective contraceptive methods (examples include oral, parenteral, or implantable hormonal contraceptive, intra-uterine device, barrier contraceptive with spermicide, partner's latex condom or vasectomy) while on study treatment and for at least twelve weeks after the last dose of the IMP.
* WCBP must have a negative serum pregnancy test within 7 days prior to first dose of the IMP.
* Male patients must agree to use a latex condom, even if they had a successful vasectomy, while on study treatment and for at least twelve weeks after the last dose of the IMP.
* Male patients must agree not to donate sperm, and female patients must agree not to donate eggs, while on study treatment and for at least 12 weeks after the last dose of the IMP.
* Availability of tumor tissue sample (either an archival specimen or a fresh biopsy material) at screening.

Key Exclusion Criteria:

* Central nervous system (CNS) metastasis.
* Active or chronic skin disorder requiring systemic therapy.
* History of Steven's Johnson's syndrome or toxic epidermal necrolysis syndrome.
* Active ocular conditions requiring treatment or close monitoring, including, but not limited to: macular degeneration, papilledema, active diabetic retinopathy with macular oedema, wet age-related macular degeneration requiring intravitreal injections, or uncontrolled glaucoma.
* Persistent toxicities from previous systemic anti-neoplastic treatments of Grade >1.
* Systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to first dose of the IMP.
* Radiotherapy to lung field at a total radiation dose of ≥20 Gy within 6 months, wide-field radiotherapy (e.g., > 30% of marrow-bearing bones) within 28 days.
* Major surgery (not including placement of vascular access device or tumor biopsies) within 28 days prior to first dose of the IMP, or no recovery from side effects of such intervention.
* Significant cardiac disease, such as recent (within six months prior to first dose of the IMP) myocardial infarction or acute coronary syndromes (including unstable angina pectoris), congestive heart failure (New York Heart Association class III or IV), uncontrolled hypertension, uncontrolled cardiac arrhythmias.
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or current ILD/pneumonitis, or suspected ILD/pneumonitis (e.g., idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, etc.).
* History of thromboembolic or cerebrovascular events, including transient ischemic attacks, cerebrovascular accidents, deep vein thrombosis, or pulmonary emboli within six months prior to first dose of the IMP.
* Acute and/or clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV).
* Administration of a live vaccine within 28 days prior to the administration of the first dose of the IMP.
* Patients requiring concurrent treatment of strong inhibitors or inducers of cytochrome P450 3A4 or 1A2 enzyme (CYP3A4 or CYP1A2) within 2 weeks prior to the first dose and during the study treatment.
* Patient who has active graft versus host disease, or diagnosis of immunodeficiency, or has an active autoimmune disease or other conditions that require systemic steroid therapy, i.e. > 10 mg daily prednisone equivalents within 14 days prior to the administration of the first dose; the use of short-course systemic corticosteroids (≤ 7 days) is permitted, with a wash-out period of 1 week prior to the administration of the first dose of the IMP.
* Known or suspected severe allergy/hypersensitivity (resulting in treatment discontinuation) to monoclonal antibodies.
* Known or suspected intolerance to the components of the IMP.
* Concurrent participation in another investigational therapeutic clinical trial.
* Patients with known active alcohol or drug abuse.
* Pregnant or breast-feeding females.
* Mental or medical conditions that prevent the patient from giving informed consent or complying with the trial or other severe acute or chronic medical or psychiatric conditions or laboratory abnormality that may increase the risk associated with the study participation or the IMP administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for enrolment in this study.
* Prior history of malignancy other than inclusion diagnosis within five years prior to first dose of the IMP.

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 24 months
  The RP2D will be determined using dose limiting toxicities (DLTs) and all other available study data
Maximum Tolerated Dose (MTD) | Up to 24 months
  The MTD will be determined using DLTs
Type, incidence and severity of Adverse Events | Up to 24 months
  Safety and tolerability profile assessed by the Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Overall Response Rate (ORR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 24 months
  Proportion of patients achieving Complete Response (CR) or Partial Response (PR)
Disease Control Rate (DCR) according to the RECIST v1.1 | Up to 24 months
  Proportion of patients achieving CR, PR or Stable Disease (SD)
Progression-free Survival (PFS) | Up to 24 months
  Time from date of start of treatment to date of the first progression or death, whichever occurs first.
Concentration of anti-drug antibodies (ADA) | Up to 24 months
  Immunogenicity profile characterized by concentration of ADAs
Maximum observed concentration (C[max]) | Up to 24 months
  Pharmacokinetic profile characterized by the maximum observed concentration (C[max]) of AMT-253
Area under the curve (AUC) | Up to 24 months
  Pharmacokinetic profile characterized by the area under the curve (AUC) of AMT-253
Terminal half-life (t[1/2]) | Up to 24 months
  Pharmacokinetic profile characterized by the terminal half-life (t[1/2]) of AMT-253
Time to maximum concentration (Tmax) | Up to 24 months
  Pharmacokinetic profile characterized by the time to maximum concentration (Tmax) of AMT-253

CONTACTS AND LOCATIONS:
Locations (7):
- Australia (7):
  - Blacktown, Sydney, New South Wales
  - Chris O'Brien Lifehouse, Sydney, New South Wales
  - Maquarie University Hospital, Sydney, New South Wales
  - ICON Cancer Centre, Brisbane, Queensland
  - Southern Oncology Clinical Research, Adelaide, South Australia
  - Cabrini Malvern Hospital, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria